CLINICAL TRIAL: NCT04670432
Title: Resolution Enhancement by a Supplemental Obstruction Lessening Venoactive Drug for Eight Weeks in Deep Vein Thrombosis: A Pilot Study to Evaluate if Hydroxyethylrutoside Reduces the Risk of Post-Thrombotic Syndrome in Patients With DVT.
Brief Title: Resolution Enhancement by a Supplemental Obstruction Lessening Venoactive Drug for Eight Weeks in Deep Vein Thrombosis
Acronym: Resolve-DVT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Netherlands Thrombosis Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NL73142.068.20
Record Dates: First submitted 2020-11-20; First posted 2020-12-17 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Deep Vein Thrombosis
Keywords: Venoactive drugs; Hydroxyethylrutoside; Venoruton; Thrombus resolution; Residual Vein Obstruction; Post-Thrombotic Syndrome
MeSH Terms: conditions — Venous Thrombosis; Postthrombotic Syndrome | interventions — Hydroxyethylrutoside; troxerutin

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: While patients are aware of their treatment allocation, the physicians (incl. radiologist) and researchers are not, as to provide unbiased outcome assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Hydroxyethylrutoside oral tablet twice daily for 8 weeks starting at the time of randomization, in addition to usual care.
  Interventions: Drug: Hydroxyethylrutoside
- Control group (No Intervention): Usual care, consisting of anticoagulant treatment and elastic compression therapy for full study duration.

INTERVENTIONS:
Drug: Hydroxyethylrutoside — 500 mg film-coated tablet
  Other Names: Venoruton
  Arms: Treatment group

SUMMARY:
The RESOLVE-DVT study is a randomized single-center pilot study to determine the effects of hydroxyethylrutoside (Venoruton) on aspects of deep vein thrombosis (DVT) resolution associated with post-thrombotic syndrome (PTS). Based on these results, the investigators will estimate its potential as a preventive therapy for PTS.

Eligible consenting patients who develop an acute, objectively confirmed DVT will be randomized and equally allocated to two trial arms, either the treatment group (Venoruton tablet 500 mg twice daily) or the control group (usual care). The pilot trial consists of 5 study contacts over 12 weeks at which outcome assessment is performed: inclusion, 1 week, 4 weeks, 8 weeks, 12 weeks. Treatment allocation is masked for outcome assessors, but not for patients.

DETAILED DESCRIPTION:
Rationale: After a DVT, one in three patients develops PTS of the affected leg, despite anticoagulant treatment and elastic compression therapy (ECT) in the acute phase of DVT. Considering the major societal burden associated with PTS, supplementation of current prevention with an effective pharmacotherapeutic therapy would be of high value. Since the pathogenesis of PTS is mediated through persistent inflammation during thrombus resolution, causing damage to the vein wall resulting in venous insufficiency, the venoactive flavonoids with their vasoprotective and anti-inflammatory properties provide an excellent candidate. As investigational medicinal product, the highly effective flavonoid Hydroxyethylrutoside (Venoruton) was chosen.

Objective: To assess the effect of Venoruton on PTS-associated aspects of DVT resolution.

Study design: A single-center, randomized, controlled, pilot study.

Study population: Adults presenting themselves at the emergency department (ED) with a first, acute, proximal DVT of the lower extremity. Inclusion will be performed within 48 hours after diagnosis of DVT.

Intervention: Administration of 500 mg Venoruton twice daily for 8 weeks following DVT, in addition to standard treatment by ECT and anticoagulant therapy.

Baseline characteristics: Assessments include demographic data, smoking status, site and extension of DVT, side of affected leg, duration of complaints at time of diagnosis, risk factors for DVT (immobilisation, trauma, etc.), type of ECT, presence/suspicion of pulmonary embolism, concomitant medications.

Main study parameters: The primary study outcome is residual vein obstruction (RVO), assessed by duplex ultrasound (DUS) at 12 weeks after DVT. Main secondary outcomes are levels of circulating biomarkers and severity of PTS-characterizing clinical signs at baseline, 1 week, 4 weeks, 8 weeks and 12 weeks. Moreover, we measure quality of life (QoL) and PTS-characterizing symptoms at baseline, 4 weeks and 12 weeks.

Additional study parameters: Medication adherence and ECT compliance at 1 week, 4 weeks, 8 weeks and 12 weeks. Pill count of Venoruton at 8 weeks. Pill count of direct oral anticoagulant (DOAC) at 12 weeks. The occurrence of relevant (serious) adverse events is assessed at all visits.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Patients have a follow-up duration of 12 weeks after diagnosis of DVT. In addition to their visit at the ED, patients will visit the outpatient clinic four times during follow-up. At each visit secondary outcomes are measured through questionnaires, blood withdrawal and assessment of the affected leg. The first visit coincides with inclusion and two subsequent visits (4 and 12 weeks) coincide with the regular clinical care pathway. The primary outcome, RVO, is measured at 12 weeks after DVT by DUS. Patients allocated to the intervention group will take two oral tablets daily over a period of eight weeks. Venoruton has been established as safe with rarely occurring, mild, reversible side-effects through many years of experience.

Masking: while patients are aware of their treatment allocation, the physicians and researchers are not, as to provide unbiased outcome assessment.

ELIGIBILITY:
Inclusion Criteria:

* Adult, defined as ≥ 18 years of age
* Objectively confirmed DVT by DUS
* Proximal DVT, defined as iliofemoropopliteal venous thrombosis
* Acute DVT, defined as having symptoms for ≤ 7 days at presentation
* Willing and able to give written informed consent

Exclusion Criteria:

* Previous DVT
* Bilateral DVT
* Pre-existent chronic venous insufficiency (CEAP-criteria C ≥ 3)
* Active malignancy, inflammatory disease (e.g. rheumatoid arthritis), or immunosuppressive therapy
* Current pregnancy or breast feeding
* Indication for therapeutic thrombolysis
* Contra-indication for DOAC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
Residual Vein Obstruction | At 12 weeks
  Transversal vein diameter ≥2mm on duplex-ultrasound during full compression, which is assessed by a radiologist blinded for study allocation. A secondary assessment based on acquired images will be performed by an independent expert radiologist, again blinded for study allocation.

SECONDARY OUTCOMES:
Levels of circulating biomarkers | At time of inclusion, 1 week, 4 weeks, 8 weeks and 12 weeks
  A panel of biomarkers, associated with RVO and PTS, will be measured in venous blood at several time-points. These include markers of inflammation (e.g. IL6, IL10), cell adhesion (e.g. ICAM1, P-selectin), and remodelling (e.g. MMPs). Differences for each individual biomarker over time will be compared between groups.
Clinical sign severity | At time of inclusion, 1 week, 4 weeks, 8 weeks and 12 weeks
  Objective Villalta score + circumference calf and ankle, which is measured by an assessor blinded to study allocation. Compared to the contralateral unaffected leg.
Symptom severity | At time of inclusion, 4 weeks and 12 weeks
  Subjective Villalta score, which is answered directly by the patient through a survey
VEINS Quality of Life/Symptoms (VEINES-QOL/Sym) | At time of inclusion, 4 weeks and 12 weeks
  This disease-specific quality of life score is answered directly by the patient through a survey.
Short Form 36 Health Survey (SF-36) | At time of inclusion, 4 weeks and 12 weeks
  This general quality of life score is answered directly by the patient through a survey.
Euro Quality of Life 5D (EQ-5D) | At time of inclusion, 4 weeks and 12 weeks
  This general quality of life score is answered directly by the patient through a survey.

OTHER OUTCOMES:
Medication adherence | At 1 week, 4 weeks, 8 weeks and 12 weeks
  Using a medication adherence score, which is answered directly by the patient.
Adherence to elastic compression therapy | At 1 week, 4 weeks, 8 weeks and 12 weeks
  Question regarding frequency of use and reason for deviation, which are answered directly by the patient.
Pill counts Venoruton | At 8 weeks, which is the end of Venoruton treatment
  In patients allocated to the intervention group, an unblinded assessor will perform a pill count of Venoruton tablets, which will be compared to the amount of tablets that should have been administered.
Pill count of DOAC | At 12 weeks
  In all patients, a pill count of the DOAC tablets will be performed and compared to the total amount of tablets that should have been administered.
(Serious) adverse events | At inclusion, 1 week, 4 weeks, 8 weeks and 12 weeks.
  The occurrence of relevant (serious) adverse events is assessed at all visits.

CONTACTS AND LOCATIONS:
Overall Officials: Arina J ten Cate - Hoek, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ten Cate-Hoek AJ, Henke PK, Wakefield TW. The post thrombotic syndrome: Ignore it and it will come back to bite you. Blood Rev. 2016 Mar;30(2):131-7. doi: 10.1016/j.blre.2015.09.002. Epub 2015 Oct 9. PMID 26462885